CLINICAL TRIAL: NCT01289743
Title: An Open-label Study of Etanercept (Enbrel) Efficacy in Ankylosing Spondylitis
Brief Title: Etanercept (Enbrel) in Ankylosing Spondylitis
Acronym: Enbrel_AS-2
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: Rheumazentrum Ruhrgebiet (Other)
Responsible Party: Prof. Dr. Jürgen Braun, Herne, Prof. Dr. Joachim Sieper, Berlin, Charité, Campus Benjamin Franklin, Hindenburgdamm 30. 12203 Berlin
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Enbrel _AS-2; 202-04 (Other: Ethical Commission)
Record Dates: First submitted 2011-02-01; First posted 2011-02-04 (Estimated); Last update posted 2011-02-04 (Estimated); Status verified 2002-02

CONDITIONS: Ankylosing Spondylitis
Keywords: ankylosing spondylitis; atanercept; therapy; magnetic resonance imaging
MeSH Terms: conditions — Spondylitis, Ankylosing | interventions — Etanercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Etanercept 25 mg (Experimental): Etanercept 25 mg subcutaneously twice weekly
  Interventions: Drug: Etanercept

INTERVENTIONS:
Drug: Etanercept — Etanercept 25 mg subcutaneously twice a week
  Other Names: Enbrel

SUMMARY:
The study has the aim to investigate the efficacy and safety of etanercept in patients with active ankylosing spondylitis (AS) over 520 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Patients 18 to 65 years of age.
2. Proven ankylosing spondylitis according to the modified New York criteria
3. Acute phase of disease with high disease activity the Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) score ≥ 4 or a pain score ≥ 4 on a Numeric Rating Scale (NRS) at two occasions in 2 weeks
4. Understand, sign. and date the written informed consent at the screening visit.
5. Sexually active women participatittg in the study must use a medically acceptable form of contraception until 6 month after the last injection of study medication. Medically acceptable forms of contraception include oral contraceptives, injectable or implantable methods, intrauterine devices, or properly used barrier contraception. Additionally, the use of condoms is suggested as an adjunct to the methods previously addressed to protect against sexually transmitted diseases and to provide additional protection against accidental pregnancy.
6. Sexually active men must agree to use a medically accepted form of contraception during the study until 6 month after the last injection of study medication.
7. Negative serum or urine pregnancy test taken at screen in all women except those surgically sterile or at least 1 year postmenopausal.
8. Able to self-administer injectable drug supplies or have a caregiver who will do so.
9. Able to store injectable test article at 2° to 8° C.

Exclusion Criteria:

1. Pregnancy/lactation
2. Previously exposure to murine or chimeric monoclonal antibodies
3. Receipt of any live (attenuated) vaccines within 4 weeks before screening visit
4. History of chronic or a recent serious infection
5. History of tuberculosis within the last 3 years
6. History of malignancy
7. Significant concurrent medical diseases including uncompensated congestive heart failure, myocardial infarction within 12 months, stable or unstable angina pectoris, uncontrolled hypertension, severe pulmonary disease, history of human immunodeficiency virus (HIV) infection, central nervous system demyelinating events suggestive of multiple sclerosis
8. Presence or history of confirmed blood dyscrasias
9. History of any viral hepatitis within 1 year prior screening or history of any drug-induced liver injury at any time prior to screening
10. Laboratory exclusions are: hemoglobin level < 8,5 mg/dl white blood cell count < 3.5 x 10^9/l platelet count < 125 x 10^9 /l creatinine level > 175 mcmol/l, liver enzymes > 1.5 times the upper limit of normal or alkaline phosphatase > 2 times the upper limit of normal.
11. Participation in trials of other investigational medications within 30 days of entering the study
12. Clinical examination showing significant abnormalities of clinical relevance
13. Concomitant medication with disease-modifying anti-rheumatic drugs (DMARDs) or corticosteroids
14. History or current evidence of abuse of "hard" drugs (eg., cocaine/heroine) or alcoholism

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2002-02; Primary Completion 2003-09 (Actual); Study Completion 2012-05 (Estimated)

PRIMARY OUTCOMES:
The Bath Ankylosing Spondylitis Disease Activity Index (BASDAI)50 response | at week 12
  Achievement of at least 50% improvement of the Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) at week 12 as compared to baseline

SECONDARY OUTCOMES:
Sustained response | every 3 months througout the study
  Percentage of patients achieving the BASDAI50 response over time
Safety outcome | at 6 and 12 weeks, every 12 weeks thereafter
  Percentage of patients experienced adverse event during the study
Magnetic resonance imaging (MRI) response | at week 24, 54, 102, 210, 308, 416, 514
  Reduction of inflammation seen on MRI in comparison to baseline
X-ray progression | at week 54, 102, 210, 308, 514
  Progression of the spinal structural changes as assessed by x-ray in comparison to baseline

CONTACTS AND LOCATIONS:
Overall Officials: Joachim Sieper, Prof. Dr., Principal Investigator — Charite University, Berlin, Germany
Locations (2):
- Germany (2):
  - Charite Campus Benjamin Franklin, Rheumatology, Berlin
  - Rheumazentrum Ruhrgebiet, Herne

REFERENCES:
- [Derived] Baraliakos X, Haibel H, Fritz C, Listing J, Heldmann F, Braun J, Sieper J. Long-term outcome of patients with active ankylosing spondylitis with etanercept-sustained efficacy and safety after seven years. Arthritis Res Ther. 2013;15(3):R67. doi: 10.1186/ar4244. PMID 23786760